CLINICAL TRIAL: NCT01701986
Title: Gemcitabine/Clofarabine/Busulfan and Allogeneic Transplantation for Aggressive Lymphomas
Brief Title: Gemcitabine Hydrochloride, Clofarabine, and Busulfan Before Donor Stem Cell Transplant in Treating Patients With Refractory B-Cell or T-Cell Non-Hodgkin Lymphoma or Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0506; NCI-2012-02055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0506 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hematopoietic Cell Transplantation Recipient; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Refractory T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Hodgkin Disease; Lymphoma, T-Cell | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Clofarabine; Gemcitabine; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Rituximab; CT-P10; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (gemcitabine, clofarabine, busulfan, BMT or PBSCT) (Experimental): PREPARATIVE REGIMEN: Patients receive gemcitabine hydrochloride IV over 40-180 minutes on days -6 and -4, clofarabine IV over 1 hour on days -6 to -3, and busulfan IV over 3 hours on days -6 to -3. Patients with matched unrelated donors also receive antithymocyte globulin IV on days -3 to -1 and patients with CD20-positive disease also receive rituximab IV on days -14, -7, 1, and 8.
  TRANSPLANT: Patients undergo allogeneic BMT or PBSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously over 24 hours or PO beginning on day -2 for up to 6 months and mycophenolate mofetil IV over 2 hours or PO TID beginning day 0.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Busulfan; Drug: Clofarabine; Drug: Gemcitabine Hydrochloride; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Biological: Rituximab; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic BMT
  Other Names: Allo BMT; Allogeneic BMT
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic BMT or PBSCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Drug: Mycophenolate Mofetil — Given IV then PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Tacrolimus — Given IV then PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase I/II trial studies the side effects and best dose of gemcitabine hydrochloride, clofarabine, and busulfan before donor stem cell transplant and to see how well it works in treating patients with B-cell or T-cell non-Hodgkin lymphoma or Hodgkin lymphoma that does not respond to treatment. Giving chemotherapy before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) of infusional gemcitabine (gemcitabine hydrochloride) combined with fixed doses of clofarabine and busulfan in patients with lymphoma receiving an allogeneic stem-cell transplant (alloSCT).

II. To estimate the day +100 success rate, defined as percentage of patients who are alive, engrafted and without grade 3-4 graft-versus (vs.)-host-disease (GVHD).

SECONDARY OBJECTIVES:

I. To estimate the day +100 success rate (defined as percentage of patients who are alive, engrafted and without grade 3-4 graft-vs.-host-disease [GVHD]).

II. To estimate the rate of event-free (EFS). III. To estimate the rate of overall survival (OS). IV. To estimate the response rate (RR) (defined as # of responses / # of patients with measurable tumors).

V. To estimate the complete response (CR) rate (defined as # of complete responses / # of patients with measurable tumors).

VI. To estimate the incidence of grade 2-4 and grade 3-4 acute GVHD. VII. To estimate the incidence of limited and extensive chronic GVHD.

OUTLINE: This is a phase I, dose-escalation study of gemcitabine hydrochloride followed by a phase II study.

PREPARATIVE REGIMEN: Patients receive gemcitabine hydrochloride intravenously (IV) over 40-180 minutes on days -6 and -4, clofarabine IV over 1 hour on days -6 to -3, and busulfan IV over 3 hours on days -6 to -3. Patients with matched unrelated donors also receive antithymocyte globulin IV on days -3 to -1 and patients with cluster of differentiation (CD)20-positive disease also receive rituximab IV on days -14, -7, 1, and 8.

TRANSPLANT: Patients undergo allogeneic bone marrow (BMT) or peripheral blood stem cell transplant (PBSCT) on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously over 24 hours or orally (PO). Beginning on day 0, patients receive mycophenolate mofetil IV over 2 hours or PO thrice daily (TID).

After completion of study treatment, patients are followed up at 3, 6, and 12 months, and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory B-cell or T-cell non-Hodgkin's lymphoma or Hodgkin's lymphoma who are eligible for allogeneic transplantation
* An 8/8 human leukocyte antigen (HLA) matched (high resolution typing at A, B, C, DRB1) sibling or unrelated donor
* Left ventricular ejection fraction (EF) >= 45%
* Forced expiratory volume in one second (FEV1) >= 50%
* Forced vital capacity (FVC) >= 50%
* Diffusing capacity of the lung for carbon monoxide (DLCO) >= 50%
* Estimated serum creatinine clearance >= 50 ml/min (using the Cockcroft-Gault formula)
* Serum creatinine =< 1.6 mg/dL
* Serum bilirubin =< 2 x upper limit of normal
* Serum glutamate pyruvate transaminase (SGPT) =< 2 x upper limit of normal
* Voluntary signed Institutional Review Board (IRB)-approved informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study; female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study; male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Patient with active central nervous system (CNS) disease
* Pregnancy (positive beta human chorionic gonadotropin [HCG] test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization) or currently breast-feeding; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Active hepatitis B, either active carrier (hepatitis B virus surface antigen [HBsAg] +) or viremic (hepatitis B virus [HBV] deoxyribonucleic acid [DNA] >= 10,000 copies/mL, or >= 2,000 IU/mL)
* Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology
* Human immunodeficiency virus (HIV) infection
* Active uncontrolled bacterial, viral or fungal infections
* Exposure to other investigational drugs within 2 weeks before enrollment
* Grade >= 3 non-hematologic toxicity from previous therapy that has not resolved to =< grade 1
* Radiation therapy to head and neck (excluding eyes), and internal organs of chest, abdomen or pelvis in the month prior to enrollment
* Prior whole brain irradiation
* Prior autologous stem-cell transplant (SCT) in the prior 3 months

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-10-25 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago L Nieto, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in MD Anderson Cancer Center
Groups:
- Cohort 1_475mgm2; Cohort 2_675mgm2; Cohort 3_975mgm2: PREPARATIVE REGIMEN: Patients receive gemcitabine hydrochloride IV over 40-180 minutes on days -6 and -4, clofarabine IV over 1 hour on days -6 to -3, and busulfan IV over 3 hours on days -6 to -3. Patients with matched unrelated donors also receive antithymocyte globulin IV on days -3 to -1 and patients with CD20-positive disease also receive rituximab IV on days -14, -7, 1, and 8.
  TRANSPLANT: Patients undergo allogeneic BMT or PBSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously over 24 hours or PO beginning on day -2 for up to 6 months and mycophenolate mofetil IV over 2 hours or PO TID beginning day 0.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic BMT
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic BMT or PBSCT
  Anti-Thymocyte Globulin: Given IV
  Busulfan: Given IV
  Clofarabine: Given IV
  Gemcitabine Hydrochloride: Given IV
  Mycophenolate Mofetil: Given IV then PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSCT
  Pharmacological Study: Correlative studies
  Rituximab: Given IV
  Tacrolimus: Given IV then PO
Period: Overall Study
Arm/Group | Cohort 1_475mgm2 | Cohort 2_675mgm2 | Cohort 3_975mgm2
Started | 8 | 24 | 32
Completed | 8 | 24 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1_475mgm2 | Cohort 2_675mgm2 | Cohort 3_975mgm2 | Total
Number analyzed (Participants) | 8 | 24 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 8 | 23 | 32 | 63
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 9 | 21
  Male | 6 | 14 | 23 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 9 | 15
  Not Hispanic or Latino | 7 | 19 | 23 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 24 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Optimal Dose of Gemcitabine Hydrochloride Determined by Dose Limiting Toxicity
Description: Dose limiting toxicity is defined as number of participants experienced grade 3-4 mucositis lasting for more than 3 days at peak severity, grade 3-4 skin toxicity lasting for more than 3 days at peak severity, occurring within 30 days from transplant, or grade 4 nonhematological/noninfectious toxicity.
Time Frame: Within 30 days of transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_475mgm2 | Cohort 2_675mgm2 | Cohort 3_975mgm2
Number analyzed (Participants) | 8 | 24 | 32
Participants
  Mucositis | 0 | 6 | 20
  Skin | 0 | 0 | 0
  Nonhematological/noninfectious toxicity | 3 | 6 | 10

2. Primary Outcome: Number of Participants That Had 100 Day Success Rate Post Transplant
Description: Number of participants that are alive, engrafted, without grade 3-4 GVHD within 100 days post transplant.
Time Frame: 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_475mgm2 | Cohort 2_675mgm2 | Cohort 3_975mgm2
Number analyzed (Participants) | 8 | 24 | 32
Participants | 6 | 17 | 21

3. Secondary Outcome: Overall Survival
Description: Number of participants that are still alive 5 years post transplant.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_475mgm2 | Cohort 2_675mgm2 | Cohort 3_975mgm2
Number analyzed (Participants) | 8 | 24 | 32
Participants | 2 | 8 | 14

4. Secondary Outcome: Treatment Related Mortality
Description: Number of participants that expired from transplant other than disease relapse within the first 100 days post transplant.
Time Frame: Up to 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_475mgm2 | Cohort 2_675mgm2 | Cohort 3_975mgm2
Number analyzed (Participants) | 8 | 24 | 32
Participants | 2 | 1 | 3

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Cohort 1_475mgm2 | Cohort 2_675mgm2 | Cohort 3_975mgm2
All-Cause Mortality (participants affected / at risk) | 6/8 | 16/24 | 18/32
Serious Adverse Events (participants affected / at risk) | 2/8 | 2/24 | 9/32
Other Adverse Events (participants affected / at risk) | 8/8 | 24/24 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1_475mgm2 (N=8) | Cohort 2_675mgm2 (N=24) | Cohort 3_975mgm2 (N=32)
ALT increased (Investigations) | 0 (0) | 0 (0) | 5 (5)
AST increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Bacterial (Infections and infestations) | 1 (1) | 2 (2) | 9 (9)
BL OTH (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Broncholitis obliterans (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
GI OTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhagic Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Low granulocyte (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Low platelet (Investigations) | 0 (0) | 0 (0) | 4 (4)
Other (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Primary graft failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Secondary graft failure (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Sepsis like syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Viral (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1_475mgm2 (N=8) | Cohort 2_675mgm2 (N=24) | Cohort 3_975mgm2 (N=32)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ALK increased (Investigations) | 1 (1) | 2 (2) | 11 (11)
ALT increased (Investigations) | 7 (7) | 16 (16) | 32 (34)
Anemia (Investigations) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ascitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
AST increased (Investigations) | 0 (0) | 4 (4) | 17 (17)
Bacterial (Infections and infestations) | 7 (7) | 24 (31) | 32 (46)
Bleeding (no GI no PUL) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Broncholitis obliterans (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic GVHD (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 5 (5) | 12 (12)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 15 (15) | 28 (28)
Dry eye (Eye disorders) | 3 (3) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Ejection fraction decreased (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 16 (16) | 24 (24)
Fever (General disorders) | 3 (3) | 8 (8) | 11 (11)
Flu like syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (General disorders) | 5 (5) | 13 (13) | 22 (22)
Fungal (Infections and infestations) | 1 (1) | 6 (6) | 3 (3)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
GI OTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
GI ULC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haptoglobin (Investigations) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 6 (6)
Hemorrhagic Cystitis (Renal and urinary disorders) | 0 (0) | 5 (5) | 11 (11)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
HP OTH (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 6 (6) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
LDH increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Low granulocyte (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Low platelet (Investigations) | 0 (0) | 0 (0) | 0 (0)
Lower Gl track obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 24 (31) | 32 (52)
Ocular GvHD (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Oral GvHD (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Oral mucositis (Gastrointestinal disorders) | 8 (8) | 24 (26) | 32 (34)
Other (General disorders) | 0 (0) | 0 (0) | 3 (3)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (5)
Parasite (Infections and infestations) | 1 (1) | 1 (1) | 5 (5)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 5 (5)
PRES (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
PU OTH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 17 (17) | 5 (5)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 5 (5)
Schistocytes (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
Serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 5 (5)
T bilirubin increased (Investigations) | 6 (6) | 15 (15) | 5 (5)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (3) | 5 (5)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Viral (Infections and infestations) | 7 (7) | 24 (34) | 32 (45)
VOD (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wbc decreased (Investigations) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT01701986/Prot_SAP_000.pdf